CLINICAL TRIAL: NCT05999019
Title: Appraisal of Surgical Outcomes and Oncological Efficiency of Intraoperative Adverse Events in Robotic Radical Gastrectomy for Gastric Cancer
Brief Title: Intraoperative Adverse Events in Robotic Radical Gastrectomy for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Other Study IDs: RGiAE-01
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: robotic surgery — robotic surgery

SUMMARY:
Surgical quality control is a crucial determinant of evaluating the tumor efficacy. We assess the ClassIntra grade for quality control and oncological outcomes of robotic radical surgery for gastric cancer (GC).

DETAILED DESCRIPTION:
Gastric cancer (GC) is the fifth most common malignant tumor worldwide and the fourth leading cause of cancer-related deaths. Surgery remains the cornerstone of GC treatment, and there is a significant lack of research on iAE compared with postoperative complications. Owing to the influence of reporting and cultural acceptance, there have been issues of inadequate reporting and non-standardized practices regarding iAE reporting.

The previously reported laparoscopic results showed that the ClassIntra grade is an effective prognostic and surgical quality control index for laparoscopic radical surgery for gastric cancer therefore it could be included in routine hospital care and surgical quality control. (DOI: 10.1097/SLA.0000000000005727). Here, iAEs in patients who underwent robotic radical gastrectomy significantly correlated with the occurrence of postoperative complications and a poor long-term prognosis. Therefore, utilization and inclusion of ClassIntra grading as a crucial surgical quality control and prognostic indicator in the routine surgical quality evaluation system are recommended.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastric adenocarcinoma through pathology;
* Preoperative chest radiograph, abdominal ultrasonogram, and full abdominal CT examination showed no distant metastasis to the liver, lungs, or abdominal cavity;
* Patients who underwent robotic radical gastrectomy.

Exclusion Criteria:

* Intraoperatively existing distant metastases
* Neoadjuvant chemotherapy
* Missing general and video data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included 366 patients who underwent robotic gastrectomy at the Department of Gastrointestinal Surgery, Fujian Medical University Union Hospital, between August 2016 and September 2019, where over 800 gastrectomies were performed annually for patients with GC.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
ClassIntra grade | 1 months
  Patients who experienced iAE were classified into the iAE group using ClassIntra grading (version 1.0). The iAEs were further classified into five sublevels (ranging from I to V according to severity) based on the ClassIntra grade

SECONDARY OUTCOMES:
Objective Structured Assessment of Technical Skill (OSATS) | 1 months
  Surgical performance was assessed using the Objective Structured Assessment of Technical Skill (OSATS)
3-year overall survival | 36 months
  Overall survival (OS) was calculated from the date of surgery to death from any cause or the last follow-up.
3-year disease-free survival | 36 months
  Disease-free survival (DFS) was calculated from the date of surgery to recurrence (locoregional and systemic), death from any cause, or the last follow-up.